CLINICAL TRIAL: NCT04726631
Title: Insulin Analogue Versus Conventional Premixed Insulin in the Treatment of Diabetes Mellitus With Pregnancy: A Prospective Cohort Study
Brief Title: Insulin in Treatment of Diabetes Mellitus With Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS-PREG
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin, Short-Acting; Insulin, Isophane; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basal insulin analogue and premeal rapid acting insulin (Other)
  Interventions: Drug: Basal insulin analogue; Drug: rapid acting insulin
- Neutral Protamine Hagedorn with regular insulin (Other)
  Interventions: Drug: Neutral Protamine Hagedorn; Drug: regular insulin

INTERVENTIONS:
Drug: Basal insulin analogue — Analogue insulin is a sub-group of human insulin
  Arms: Basal insulin analogue and premeal rapid acting insulin
Drug: rapid acting insulin — Rapid acting insulins are usually taken just before or with a meal. They act very quickly to minimise the rise in blood sugar which follows eating.
  Arms: Basal insulin analogue and premeal rapid acting insulin
Drug: Neutral Protamine Hagedorn — is an intermediate-acting insulin
  Arms: Neutral Protamine Hagedorn with regular insulin
Drug: regular insulin — is a type of short-acting insulin.
  Arms: Neutral Protamine Hagedorn with regular insulin

SUMMARY:
The prevalence of diabetes melilites is rapidly increasing over years and consequently during pregnancy. In 2017, there were 21.3 million pregnant women who experienced hyperglycemia, of which 86.4% of them were diagnosed with gestational diabetes melilites.

Pregnancy in women with diabetes is associated with an intensification in adverse maternal, fetal and perinatal outcomes including spontaneous abortions, congenital malformations, preterm labor, and macrosomia. Several studies have confirmed that poor glycemic control in women with either gestational, type 1 or type 2 diabetes during pregnancy is associated with poor pregnancy outcomes. In the same line, proper glycemic control before, early, and through all pregnancy markedly improves both maternal and fetal outcomes.

Insulin therapy is the standard treatment of diabetes melilites with the pregnancy if dietary control and exercise fail. However, insulin therapy has its difficulties like approaches to mimicking postprandial insulin release, providing adequate background insulin, balancing insulin dosage, food, activity, hypoglycemic episodes, overall glycemia. This is always a struggle for doctors and patients and much affecting their lifestyle

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 45 years old,
* Women with pre-gestational diabetes.
* Those who were under premixed insulin therapy prior to pregnancy.
* women pregnant between 14 weeks up to 28 weeks of gestation

Exclusion Criteria:

* History of recurrent miscarriage
* multiple pregnancies
* chronic hypertension
* severe heart, liver, and kidney disease.
* women how got pregnant after assisted reproduction
* those with advanced retinopathy, hypersensitivity to insulin.
* Women who developed bleeding in early pregnancy and those diagnosed to have any major anomaly during the first-trimester scan.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
the percentage of maternal glycosylated Hemoglobin | 6 months